CLINICAL TRIAL: NCT05350137
Title: Application of Carbon Dioxide for Identifying the Intersegmental Plane in Thoracoscopic Segmentectomy: A Randomized Controlled Study
Brief Title: Application of Carbon Dioxide for Identifying the Intersegmental Plane in Thoracoscopic Segmentectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhang Ni, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TJ-IRB20220140
Record Dates: First submitted 2022-02-16; First posted 2022-04-27 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer; Pulmonary Nodule, Solitary; Segmentectomy; Pulmonary Nodule, Multiple
Keywords: Lung segmentectomy; Intersegmental plane; Inflation-deflation method; Carbon dioxide
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule; Multiple Pulmonary Nodules | interventions — Oxygen; Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: 100% oxygen (Active Comparator): After dividing all the targeted vascular and bronchial structures, the lung of the operating side was re-inflated with 100% oxygen.
  Interventions: Procedure: 100% oxygen
- Group B: Carbon dioxide (Experimental): After the targeted segment structures were successfully dissected, the collapsed intraoperative lung was completely re-expanded with carbon dioxide.
  Interventions: Procedure: Carbon dioxide

INTERVENTIONS:
Procedure: 100% oxygen — During one-lung ventilation with an open chest, the non-ventilated lung collapses initially due to the inherent elastic recoil properties of the lung. Once passive venting has ceased, further collapse will then be wholly dependent on ongoing gaseous uptake and absorption atelectasis. Improved inflation-deflation method is currently the most widely used method in clinical practice. After dividing all the targeted vascular and bronchial structures, the lung of the operating side was re-inflated with 100% oxygen. After the operative lungs is completely expanded, perform pure oxygen mechanical single lung ventilation for the healthy lung, waiting for clear presentation of the plane between the targeted segment and the other segments.
  Arms: Group A: 100% oxygen
Procedure: Carbon dioxide — During one-lung ventilation with an open chest, the non-ventilated lung collapses initially due to the inherent elastic recoil properties of the lung. Once passive venting has ceased, further collapse will then be wholly dependent on ongoing gaseous uptake and absorption atelectasis. The solubility coefficient for carbon dioxide is 0.57. The rapid diffusion properties of carbon dioxide would be expected to speed lung collapse and so facilitate surgery. After the targeted segment structures were successfully dissected, the collapsed intraoperative lung was completely re-expanded with carbon dioxide. After the operative lungs is completely expanded, perform pure oxygen mechanical single lung ventilation for the healthy lung, waiting for clear presentation of the plane between the targeted segment and the other segments.
  Arms: Group B: Carbon dioxide

SUMMARY:
With the increasing acceptance of routine computed tomography (CT) screenings, early-stage lung cancer detection is becoming more frequent. For ground glass opacity predominant early-stage lung cancer, segmentectomy can get the same oncological benefits as lobectomy. In addition, lung nodules that are highly suspected to be metastases can also be performed by segmentectomy to preserve more lung function. During the surgery, the rapid and precise identification of the intersegmental plane is one of the challenges. The improved inflation-deflation method is currently the most widely used method in clinical practice. According to the dispersion coefficient of the gas, the rapid diffusion properties of carbon dioxide would be expected to speed lung collapse and so facilitate surgery. The purpose of this study was to investigate the feasibility and safety of carbon dioxide on the appearance time of satisfactory and ideal planes during segmentectomy.

DETAILED DESCRIPTION:
This study was approved by the ethics committee of Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology. This randomized parallel group trial enrolled patients scheduled to receive thoracoscopic anatomic segmentectomy at Tongji Hospital. General anesthesia with double lumen endotracheal tube was administered to the patients. With the guidance of preoperative three-dimensional computed tomography bronchography and angiography, the targeted segment structures could be precisely dissected, and then intersegmental demarcation was confirmed by the modified inflation-deflation method in this study. In group A (100% oxygen), after dividing all the targeted vascular and bronchial structures, the lung of the operating side was re-inflated with 100% oxygen. In group B (Carbon dioxide), after the targeted segment structures were successfully dissected, the collapsed operative lung was completely re-expanded with carbon dioxide. The purpose of this study was to investigate the feasibility and safety of carbon dioxide on the appearance time of satisfactory and ideal planes during segmentectomy. The starting time point of the intersegmental plane was when the whole lungs had completely re-expanded. The end point was when the preserved segment was fully deflated, and a boundary had formed between the targeted segment and the reserved lung.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years of age.
2. Segmentectomy is feasible according to the reconstructed 3-dimensional (3D) images.
3. Pulmonary nodule 2 cm or smaller in diameter with 50% or more ground-glass opacity (GGO) on thin-slice computed tomography, indicating an underlying malignancy.
4. Ability to provide written informed consent.
5. Unable to tolerate lobectomy as indicated by standard clinical pre-op evaluation, including pulmonary function tests and cardiac evaluation.
6. Diagnosis confirmed or suspected of lung metastatic cancer.

Exclusion Criteria:

1. Patients who are at risk for general anesthesia.
2. Patients with serious mental illness.
3. Pregnancy or lactating women.
4. Active bacterial or fungal infections.
5. Panties with Interstitial pneumonia, pulmonary fibrosis or severe emphysema.
6. Conversion to thoracotomy in surgery.
7. Preoperative assessment of patients undergoing lobectomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A: 100% Oxygen | Group B: Carbon Dioxide
Started | 26 | 26
Completed | 23 | 18
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 100% Oxygen | Group B: Carbon Dioxide | Total
Number analyzed (Participants) | 23 | 18 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.00 (13.19) | 51.17 (12.48) | 51.07 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 23 | 18 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 23 | 18 | 41
body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.6 (2.9) | 23.8 (3.0) | 23.1 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: The Intersegmental Border Appearance Time During the Surgery.
Description: The starting time point of the intersegmental plane was when the whole lungs had completely re-expanded. The end point was when the preserved segment was fully deflated, and a boundary had formed between the targeted segment and the reserved lung.
Time Frame: The time of appearance of the intersegmental plane that can be performed satisfactorily by surgeons during the surgery.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group A: 100% Oxygen | Group B: Carbon Dioxide
Number analyzed (Participants) | 23 | 18
seconds | 748.74 (177.16) | 157.11 (76.75)

2. Secondary Outcome: The Arterial Blood Gas Results During Perioperative Period.
Description: Extracting arterial blood gas.
Time Frame: Immediately after the radial arterial catheterization when inhaling the air, pre-intervention, 3-minutes, 5-minutes, 15-minutes during the single lung ventilation after the intervention.
Reporting Status: Not Posted

3. Other Pre Specified Outcome: The Incidence of Postoperative Complications.
Description: Record the complications.
Time Frame: 4 weeks after surgery.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: The Length of Hospital Stays.
Description: Duration of hospitalization after surgery.
Time Frame: Up to 14 days.
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Quality of Recovery.
Description: Measured using the Quality of Recovery 40 (QoR-40) Score and asking patients to complete the questions 24 hours before operation, 48 hours after operation and 1 week after operation.
Time Frame: Up to 7 days.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 weeks after surgery
Arm/Group | Group A: 100% Oxygen | Group B: Carbon Dioxide
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/18
Other Adverse Events (participants affected / at risk) | 5/23 | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: 100% Oxygen (N=23) | Group B: Carbon Dioxide (N=18)
Air leakage (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT05350137/Prot_SAP_000.pdf